CLINICAL TRIAL: NCT02540122
Title: Imaging of Conjunctival Microvasculature During Contact Lens Wear
Brief Title: Pilot Clinical Evaluation of Approved Contact Lenses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5627
Record Dates: First submitted 2015-08-31; First posted 2015-09-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Subject A (Neophytes) (Active Comparator): Subjects will wear the Marketed Contact Lens 1, Marketed Contact Lens 2, Marketed Contact Lens 3, and Marketed Contact Lens 4 for a 6-hour period in a bilateral and random fashion, with a washout period of one week between lenses. Each subject will randomly be assigned to one of four unique sequences of a 4 x 4 crossover design. A block size of two sequences will be used.
  Interventions: Device: Marketed Contact Lens 1; Device: Marketed Contact Lens 2; Device: Marketed Contact Lens 3; Device: Marketed Contact Lens 4
- Subject B (Habitual Lens Wearers) (Active Comparator): Subjects will wear the Marketed Contact Lens 1, Marketed Contact Lens 2, Marketed Contact Lens 3, and Marketed Contact Lens 4 for a 6-hour period in a bilateral and random fashion, with a washout period of one week between lenses. Each subject will randomly be assigned to one of four unique sequences of a 4 x 4 crossover design. A block size of two sequences will be used.
  Interventions: Device: Marketed Contact Lens 1; Device: Marketed Contact Lens 2; Device: Marketed Contact Lens 3; Device: Marketed Contact Lens 4

INTERVENTIONS:
Device: Marketed Contact Lens 1 — Marketed contact lens being worn by the subject in a bilateral fashion for approximately 6 hours (+/- 30 minutes).
  Other Names: etafilcon A
Device: Marketed Contact Lens 2 — Marketed contact lens being worn by the subject in a bilateral fashion for approximately 6 hours (+/- 30 minutes).
  Other Names: nelfilcon A
Device: Marketed Contact Lens 3 — Marketed contact lens being worn by the subject in a bilateral fashion for approximately 6 hours (+/- 30 minutes).
  Other Names: narafilcon A in 8.5 base curve
Device: Marketed Contact Lens 4 — Marketed contact lens being worn by the subject in a bilateral fashion for approximately 6 hours (+/- 30 minutes).
  Other Names: narafilcon A in 9.0 base curve

SUMMARY:
This is a pilot evaluation to assess the feasibility of using novel imaging process to characterize lens edge and limbal epithelial thickness profile; lens movement with gaze and blink; and conjunctival microvasculature including fractal analysis of microvascular perfusion maps and blood flow velocity.

DETAILED DESCRIPTION:
This is a pilot evaluation to assess the feasibility of using ultra-high resolution optical coherence tomography (OCT) to image and characterize lens edge and limbal epithelial thickness profile; lens movement with gaze and blink; and conjunctival microvasculature including fractal analysis of microvascular perfusion maps and blood flow velocity.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 and not more than 70 years of age.
* The subject's refractive cylinder must be < 1.00 Diopters (D) in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.
* The subject must be either a neophyte or a habitual and adapted wearer of soft contact lenses in both eyes.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* The subject must demonstrate adequate mobility and 20/30 vision oculus dexter (OD) and oculus sinister (OS) with the study contact lenses.

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in-situ keratomileusis (LASIK), etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Monovision or multi-focal contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self report).
* Suspicion of or recent history of alcohol or substance abuse.
* History of serious mental illness.
* History of seizures.
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Assessment of Bulbar Conjunctival Blood Flow Velocity | 4 contact lenses will be tested over a period of 21 days.
  Bulbar conjunctival microvascular responses among different types of contact lenses after a period of lens wear will be observed and evaluated for clinical relevance findings.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States